CLINICAL TRIAL: NCT05290506
Title: Association of Fasting GLP-1 Level With the Effect of Linagliptin After an Oral Glucose Tolerance Test in Prediabetes and Type 2 Diabetes Mellitus
Brief Title: Linagliptin Response to OGTT in Prediabetes and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Chong Shiau Chin, Mrs, principal investigator, National University of Malaysia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Linagliptin study
Record Dates: First submitted 2022-02-25; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: PreDiabetes; Type 2 Diabetes
Keywords: glucagon-like peptide 1; Dipeptidyl peptidase inhibitor; oral glucose tolerance test; prediabetes; type 2 diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors; Linagliptin

STUDY DESIGN:
Intervention Model Description: open-labelled, single treatment study between Low GLP-1 group and High GLP-1 group of prediabetes/type 2 diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prediabetes Low GLP-1 (Active Comparator): prediabetes patients were divided into high GLP-1 and low GLP-1 groups based on the median of fasting GLP-1 level. linagliptin 5mg once daily was administered.
  Interventions: Drug: Dipeptidyl-Peptidase IV Inhibitors
- Prediabetes High GLP-1 (Active Comparator): prediabetes patients were divided into high GLP-1 and low GLP-1 groups based on the median of fasting GLP-1 level. linagliptin 5mg once daily was administered.
  Interventions: Drug: Dipeptidyl-Peptidase IV Inhibitors
- Diabetes Low GLP-1 (Active Comparator): type 2 diabetes mellitus patients were divided into high GLP-1 and low GLP-1 groups based on the median of fasting GLP-1 level. linagliptin 5mg once daily was administered.
  Interventions: Drug: Dipeptidyl-Peptidase IV Inhibitors
- Diabetes High GLP-1 (Active Comparator): type 2 diabetes mellitus patients were divided into high GLP-1 and low GLP-1 groups based on the median of fasting GLP-1 level. linagliptin 5mg once daily was administered.
  Interventions: Drug: Dipeptidyl-Peptidase IV Inhibitors

INTERVENTIONS:
Drug: Dipeptidyl-Peptidase IV Inhibitors — All subjects were given linagliptin 5mg once daily for 12 weeks. Comparison of their OGTT response at week 0 and week 12
  Other Names: linagliptin

SUMMARY:
There are studies that suggest glycemic response to incretin-based therapies differs between Asians and Caucasians, whereby Asians have better response compared to Caucasians. Hence, the therapeutic response could also be augmented by difference in incretin system among various ethnicities. This study is carried out to study the effect of dipeptidyl-peptidase IV (DPPIV) inhibitors in prediabetes and T2DM patients who have different levels of GLP-1 and to determine the effect on glycemic profiles, insulin resistance/sensitivity, beta-cell functon.

DETAILED DESCRIPTION:
A 12-week, open-label, single treatment study using linagliptin is conducted in 28 prediabetes and 22 T2DM subjects who are divided into low and high fasting GLP-1 groups. Prediabetes are recruited from OGTT screening. Type 2 diabetes patients are recruited from specialised diabetes clinic and routine follow-up. A 75-g oral glucose tolerance test (OGTT) is performed at week 0 and 12. Venous blood samples were drawn at times 0 (before initiation of OGTT), 30, 60, 90, 120 min from the indwelling catheter for measurement of glucose and insulin.All prediabetes and T2DM subjects receive Linagliptin 5mg once daily for a duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes diagnosed from OGTT and T2DM subjects
* HbA1c > 6.5% and <10%
* Subjects not receiving any glucose-lowering medication or just receiving metformin and/or sulphonylureas and/or alpha-glucosidase inhibitors on stable dose for at least 3 months.
* Subjects who are willing to participate and sign the informed consent form

Exclusion Criteria:

* Subjects with ketoacidosis or lactic acidosis, overt diabetes, another disease causing secondary glucose intolerance, congestive heart failure (New York Heart Association Class III or IV), myocardial infarction, stroke or ischemic attacks in past 6 months, uncontrolled severe hypertension, active liver conditions such as cirrhosis or hepatitis [elevation in liver enzymes to higher activities than double the respective normal value], moderate to severe renal insufficiency, pregnancy, breast-feeding
* Patients receiving insulin, GLP-1 receptor agonists, dipeptidyl peptidase IV inhibitors or glucose-lowering medications other than metformin /sulphonylureas /alpha-glucosidase inhibitors as treatment.
* Subjects with uncontrolled blood glucose HbA1c>10%
* Subjects who plan to move out of state / country

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in glucose after 12-week treatment | baseline to 12 weeks
  OGTT is performed at week 0 (baseline) and 12 (complete treatment). plasma glucose levels are taken at time 0,30,60,90,120 minutes during OGTT.
change from baseline in HbA1c after 12-week treatment | baseline to 12 weeks
  plasma level of fasting HbA1c is taken at week 0 and 12 of study before OGTT
change from baseline in insulin sensitivity/resistance index after 12-week treatment | baseline to 12 weeks
  OGTT is performed at week 0 (baseline) and 12. Plasma levels of glucose and insulin are taken at time 0,30,60,90,120 min during the OGTT. HOMA-IR, HOMA-IS are used to measure insulin resistance and insulin sensitivity at week 0 and week 12

SECONDARY OUTCOMES:
change from baseline in beta-cell function after 12-week treatment | baseline to 12 weeks
  OGTT is performed at week 0 (baseline) and 12 (treatment complete). HOMS-beta, insulinogenic index, oral disposition index are used to measure beta-cell funciton at week 0 and 12

CONTACTS AND LOCATIONS:
Overall Officials: SHIAU CHONG, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Sultan Ismail, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No